CLINICAL TRIAL: NCT01860417
Title: Treatment of Lumbar Degenerative Disc Disease With Allogenic Mesenchymal Stem Cells (MSV*) *MSV: Bone Marrow Mesenchymal Stromal Cells Expanded Using the Valladolid IBGM Procedure
Brief Title: Treatment of Degenerative Disc Disease With Allogenic Mesenchymal Stem Cells (MSV)
Acronym: Disc_allo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Citospin (Industry); University of Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TerCel005; 2012-004444-30 (EudraCT Number); Disc_allo_MSV (Other: Red TerCel)
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Degenerative Disc Disease; Intervertebral Disc Disease; Low Back Pain
Keywords: Degenerative Disc Disease,; Intervertebral Disc Disease; Low Back Pain; Nucleus pulposus; Stem cell; Cellular therapy; Regenerative therapy; Mesenchymal stem cells; Bone marrow; Musculoskeletal Diseases; Mesenchymal Stromal Cells (allogenic)
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease; Low Back Pain; Musculoskeletal Diseases | interventions — Genes, mos; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogenic Mesenchymal Stromal Cells (Experimental): Mesenchymal stem cells (MSC) prepared from bone marrow from healthy donor expanded ex vivo for 3-4 weeks. Intradiscal injection of 25 millions MSC in 2 ml of saline
  Interventions: Biological: Allogenic Mesenchymal Stromal Cells
- Mepivacaine (Active Comparator): Infiltration of paravertebral musculature close to the affected disc(s) with 2 ml of 1% Mepivacaine
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Biological: Allogenic Mesenchymal Stromal Cells
  Other Names: Mesenchymal stem cells (MSC); MSC injection; MSV (MSV=MSC prepared following Valladolid IBGM procedure)
  Arms: Allogenic Mesenchymal Stromal Cells
Drug: Mepivacaine
  Other Names: Sham-treated comparator; Mepivacaine is also known as Carbocaine; Mepivacaine is also known as Polocaine
  Arms: Mepivacaine

SUMMARY:
In this study we want to evaluate the clinical use of allogenic mesenchymal stem cells (MSC), obtained from bone marrow of healthy donors, for treatment of Degenerative Disc Disease (DDD). The trial is based in previous results with autologous MSC (Orozco et al., Transplantation 92: 822-828; 2011). Here we propose a phase I-II trial, prospective, randomized, blinded, and controlled for the treatment DDD using MSV, a Good Manufacturing Practice (GMP)-compliant expanded bone marrow MSC (MSV, Investigational medicinal product Num. 10-134). The assay consists of two arms with 12 patients each one. Patients in the experimental arm will be given a single intra-discal transplantation of MSV (25 millions in 2 ml). Control patients will be infiltrated in the paravertebral muscles close to the lesion with 2 ml of 1% mepivacain. We shall follow the evolution of pain, disability and quality of life as well as disc fluid content by Magnetic Resonance Imaging (T2-calibrated).

ELIGIBILITY:
Inclusion Criteria:

* Degenerative disease of one or two lumbar discs with predominant back pain after conservative treatment (physical and medical) for over 6 months.
* Fibrous ring capable of holding the cell implantation, demonstrated by Magnetic resonance imaging (MRI) image (stages 2, 3 and 4 of Adams).
* Decrease of disc height of more than 20% (radiographic measurement in side image).
* Absence of spinal infection.
* Haematological and biochemical analysis wit no significant alterations that contraindicates intervention.
* The patient is able to understand the nature of the study.
* Informed written consent of the patient.

Exclusion Criteria:

* Age over 75 or under 18 or legally dependent
* Allergy to gentamicin, or to bovine, cattle or horse serum.
* Congenital or acquired diseases leading to spine deformations that may upset cell application.
* Spinal segmental instability, spinal canal stenosis, isthmus pathology and other conditions that may compromise the study
* Modic III changes on MRI images (31).
* Overweight with body mass index (mass in Kg/size in m2) greater than 35 (obesity grade II).
* Pregnancy or breast-feeding
* Neoplasia
* Immunosuppression
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
* Other conditions that may, according to medical criteria, discourage participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Garcia-Sancho, MD, PhD, Study Chair — Scientific Park Foundation of University of Valladolid; David C Noriega, MD, PhD, Study Director — Hospital Clinico Universitario, Valladolid; Ana Sanchez, MD, PhD, Study Director — Citospin; FRancisco Ardura, MD, PhD, Principal Investigator — Hospital Clinico Universitario, Valladolid
Locations (2):
- Spain (2):
  - Hospital Clinico Universitario, Valladolid
  - Instituto de Biologia y Genetica Molecular, Valladolid

REFERENCES:
- [Background] Orozco L, Soler R, Morera C, Alberca M, Sanchez A, Garcia-Sancho J. Intervertebral disc repair by autologous mesenchymal bone marrow cells: a pilot study. Transplantation. 2011 Oct 15;92(7):822-8. doi: 10.1097/TP.0b013e3182298a15. PMID 21792091
- [Derived] Noriega DC, Ardura F, Hernandez-Ramajo R, Martin-Ferrero MA, Sanchez-Lite I, Toribio B, Alberca M, Garcia V, Moraleda JM, Sanchez A, Garcia-Sancho J. Intervertebral Disc Repair by Allogeneic Mesenchymal Bone Marrow Cells: A Randomized Controlled Trial. Transplantation. 2017 Aug;101(8):1945-1951. doi: 10.1097/TP.0000000000001484. PMID 27661661
- See also: Treatment of Degenerative Disc Disease with Autologous Mesenchymal Stem Cells — http://www.ncbi.nlm.nih.gov/pubmed/?term=orozco+and+garcia-sancho
- See also: Instituto de Biologia y Genética Molecular IBGM), Cell Production Research — http://www.ibgm.med.uva.es
- See also: Intervertebral disk — http://www.ncbi.nlm.nih.gov/mesh/?term=intervertebral
- See also: mesenchymal stem cells — http://www.ncbi.nlm.nih.gov/mesh?term=cell%2C%20mesenchymal%20stem

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed between June 2013 and March 2014. Date of Last visit last patient was December 2015. The study was conducted in only one center in Spain.
Groups:
- Allogenic Bone Marrow Mesenquimal Cells: Mesenchymal stem cells (MSC) prepared from bone marrow from healthy donor expanded ex vivo for 3-4 weeks. Intradiscal injection of 25 millions MSC in 2 ml of saline
- Mepivacaine: Infiltration of paravertebral musculature close to the affected disc(s). The control group received a sham infiltration of paravertebral musculature with the anesthetic: saline containing 1% mepivacaine (1 ml of 2% mepivacaine + 1 ml of saline).
Period: Overall Study
Arm/Group | Allogenic Bone Marrow Mesenquimal Cells | Mepivacaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 40.5 [25 to 50] | 37 [21 to 56] | 38 [21 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 11 | 22
  Hispanic | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 12 | 12 | 24
Weight [Median (Full Range); unit: Kg] | 72 [49 to 85] | 74 [46.5 to 86] | 72.5 [46.5 to 86]
Height [Median (Full Range); unit: cm] | 166.5 [150 to 191] | 176.5 [157 to 188] | 172 [150 to 191]
Body mass index [Median (Full Range); unit: kg/m^2] | 25.5 [20.9 to 31.2] | 24.0 [18.5 to 27.3] | 24.5 [18.5 to 31.2]
Participants with Previous Treatment [Count of Participants; unit: Participants] | 11 | 12 | 23
Visual Analogue Scale [Median (Full Range); unit: units on a scale] — Pain evaluation using a visual analogue scale (VAS) at baseline. Outcomes are expressed using a 0%-100% scale. A higher score indicates greater pain intensity
  units on a scale | 73.5 [31 to 100] | 72.5 [20 to 86] | 73 [20 to 100]
Oswestry Disability Index [Median (Full Range); unit: units on a scale] — Subject's Disability score in the Oswestry Disability Index (ODI) before intervention. Outcomes are expressed using a 0%-100% scale. Zero is equated with no disability and 100 is the maximum disability possible
  units on a scale | 26 [2 to 78] | 22 [4 to 46] | 24 [2 to 78]
SF-12 Physical Component [Median (Full Range); unit: units on a scale] — Results from the physical component of the short form-12 (SF-12) life quality questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
  units on a scale | 38 [28 to 53] | 42.5 [18 to 54] | 38.5 [18 to 54]
SF-12 Mental Component [Median (Full Range); unit: units on a scale] — Results from the mental component of the short form-12 (SF-12) life quality questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
  units on a scale | 50 [36 to 69] | 50 [21 to 58] | 50 [21 to 69]
Pfirrmann grading system [Count of Participants; unit: Participants] — Grades:
  * Gr I: Disc homogeneous. Bight hyperintense white signal intensity. Normal height
  * Gr II: Disc inhomogeneous. Hyperintense white signal. Nucleus/annulus clearly differentiated. Height is normal
  * Gr III: Disc inhomogeneous. Intermittent gray signal intensity. Unclear distinction nucleus/annulus. Height normal/slightly decreased
  * Gr IV: Disc inhomogeneous. Hypointense dark gray signal intensity. No distinction nucleus/annulus. Height slightly/moderately decreased.
  * Gr V: Disc inhomogeneous. Hypointense black signal intensity. No distinction nucleus/annulus. Disc space is collapsed
  Participants
    Gr II | 0 | 3 | 3
    Gr III | 5 | 8 | 13
    Gr IV | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain and Disability Evaluation
Description: Change in the composite variable, which includes pain and disability 1 year after intervention, was plotted as a function of the initial pain score or disability index. Results for the relief of lumbar pain and Oswestry disability index were all included for both, control and cell-treated patients. The scores obtained from this analysis (slope of the plot) range from 0 to 1, with higher scores meaning a better outcome.
Time Frame: Change since the baseline (before intervention) up to the end of the follow-up period, 12 months after the intervention
Measure: Mean (Standard Error); unit: scores from 0 to 1
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
scores from 0 to 1 | 0.28 (0.07) | 0.15 (0.1)

2. Secondary Outcome: Evaluation of Affected Disc(s) by Quantitative MRI Ratio 12/6months
Description: Ratio discs density: Discs density at 12 months divided by discs density at 6 months after transplantation.
  To homogenize the results of different patients, the water content values of the affected discs were normalized to the values obtained from the healthy discs in the same individual; for these purposes, the density of the affected segments was divided by the average value of the healthy discs. Finally, the value after the treatment was divided by the baseline value.
Time Frame: At 12 months from 6 months after the intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
ratio | 0.22 (0.11) | 0.06 (0.08)

3. Secondary Outcome: Evaluation of Affected Disc(s) by Quantitative Magnetic Resonance Imaging (RMI): Density at 6 Months
Description: Measurement of the amount of fluid in the disc. To homogenize the results of different patients, the water content values of the affected discs were normalized to the values obtained from the healthy discs in the same individual; for these purposes, the density of the affected segments was divided by the average value of the healthy discs. Finally, the value after the treatment was divided by the baseline value.
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
ratio | 0.42 (0.05) | 0.51 (0.05)

4. Secondary Outcome: Evaluation of Affected Disc(s) by Quantitative Magnetic Resonance Imaging (RMI): Density at 12 Months
Description: as for outcome 3
Time Frame: At 12 months after the intervention
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
ratio | 0.52 (0.06) | 0.46 (0.05)

5. Secondary Outcome: Visual Analogue Scale at 3 Months
Description: Pain evaluation using a visual analogue scale (VAS) at baseline. Outcomes are expressed using a 0%-100% scale. A higher score indicates greater pain intensity
Time Frame: At 3 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 43 (9) | 46 (8)

6. Secondary Outcome: Visual Analogue Scale at 6 Months
Description: as for outcome 5
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 40 (8) | 51 (8)

7. Secondary Outcome: Visual Analogue Scale at 12 Months
Description: as for outcome 5
Time Frame: At 12 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 47 (10) | 47 (8)

8. Secondary Outcome: Oswestry Disability Index at 3 Months
Description: Subject's Disability score in the Oswestry Disability Index (ODI) before intervention. Outcomes are expressed using a 0%-100% scale. Zero is equated with no disability and 100 is the maximum disability possible
Time Frame: At 3 months after the intervention
Measure: Mean (Standard Error); unit: percent
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
percent | 16 (6) | 25 (4)

9. Secondary Outcome: Oswestry Disability Index at 6 Months
Description: as for outcome 8
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: percent
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
percent | 20 (7) | 30 (6)

10. Secondary Outcome: Oswestry Disability Index at 12 Months
Description: as for outcome 8
Time Frame: At 12 months after the intervention
Measure: Mean (Standard Error); unit: percent
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
percent | 22 (7) | 34 (7)

11. Secondary Outcome: SF-12 Physical Component at 3 Months
Description: Results from the physical component of the short form-12 (SF-12) life quality questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Time Frame: 3 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 47 (3) | 43 (3)

12. Secondary Outcome: SF-12 Physical Component at 6 Months
Description: as for outcome 11
Time Frame: 6 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 46 (3) | 39 (3)

13. Secondary Outcome: SF-12 Physical Component at 12 Months
Description: as for outcome 11
Time Frame: 12 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 45 (3) | 42 (3)

14. Secondary Outcome: SF-12 Mental Component at 3 Months
Description: Results from the mental component of the short form-12 (SF-12) life quality questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Time Frame: 3 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 50 (2) | 46 (3)

15. Secondary Outcome: SF-12 Mental Component at 6 Months
Description: as for outcome 14
Time Frame: 6 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 52 (2) | 48 (3)

16. Secondary Outcome: SF-12 Mental Component at 12 Months
Description: as for outcome 14
Time Frame: 12 months after the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
units on a scale | 48 (3) | 50 (3)

17. Secondary Outcome: Pfirrmann Stage at 6 Months
Description: Grades:
  Gr I: Disc homogeneous. Bight hyperintense white signal intensity. Normal height Gr II: Disc inhomogeneous. Hyperintense white signal. Nucleus/annulus clearly differentiated. Height is normal Gr III: Disc inhomogeneous. Intermittent gray signal intensity. Unclear distinction nucleus/annulus. Height normal/slightly decreased Gr IV: Disc inhomogeneous. Hypointense dark gray signal intensity. No distinction nucleus/annulus. Height slightly/moderately decreased.
  Gr V: Disc inhomogeneous. Hypointense black signal intensity. No distinction nucleus/annulus. Disc space is collapsed
Time Frame: At 6 months after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 12 | 12
Participants
  Gr II | 0 | 1
  Gr III | 10 | 8
  Gr IV | 2 | 3

18. Secondary Outcome: Pfirrmann Stage at 12 Months
Description: as for outcome 17
Time Frame: At 12 months after the intervention
Population: One patient not evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
Number analyzed (Participants) | 11 | 12
Participants
  Gr II | 1 | 1
  Gr III | 9 | 4
  Gr IV | 1 | 7

ADVERSE EVENTS:
Time Frame: Adverse events reporting started when after the administration of the study treatments, and lasted up to the last visit of each patient at the end of the follow-up period, 12 months after the intervention.
Arm/Group | Allogenic Mesenchymal Stromal Cells | Mepivacaine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogenic Mesenchymal Stromal Cells (N=12) | Mepivacaine (N=12)
Device failure (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogenic Mesenchymal Stromal Cells (N=12) | Mepivacaine (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 9 (13)

LIMITATIONS AND CAVEATS:
Further studies shall track the long-term evolution as well as investigate the anatomical and functional changes that occur in the intervertebral spaces and shall increase the number of patients, which was an important limitation of the present study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-10-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT01860417/Prot_SAP_ICF_000.pdf